CLINICAL TRIAL: NCT05634694
Title: Clinical Study on the Drug Sensitivity Consistency of Patient-Derived Organoid Model and Actual Therapeutic Efficacies in Cholangiocarcinoma Patients Receiving Adjuvant Chemotherapy After Radical Resection
Brief Title: Study on Consistency Evaluation for Drug Sensitivity of Patient-Derived Organoid Model From Cholangiocarcinoma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2022-168-01
Record Dates: First submitted 2022-11-16; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Cholangiocarcinoma
Keywords: Cholangiocarcinoma; Chemotherapy; Adjuvant therapy; Patient-Derived Organoid; Drug Sensitivity
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Resected tumor samples will be used to culture organoids for drug sensitivity testing. And the organoids that are successfully cultured will be kept in liquid nitrogen for a specific time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-sen University: The cohort of Sun Yat-Sen Memorial Hospital of Sun Yat-sen University is the exploration cohort.
  Interventions: Other: No interventions.

INTERVENTIONS:
Other: No interventions. — No interventions.

SUMMARY:
This is a single-center, prospective, observational and exploratory clinical study. The object of this study is to evaluate the consistency and accuracy of patient-derived organoid model of cholangiocarcinoma to predict the clinical chemotherapeutic efficacy, as well as the possibility of guiding the adjuvant chemotherapy.

DETAILED DESCRIPTION:
The chemotherapeutic efficacy is heterogeneous among cholangiocarcinoma patients after radical resection, and an accurate and relatively convenient model evaluating the chemotherapeutic efficacy is still lacking. This study aims to prospectively evaluate the consistency of drug sensitivity between patient-derived organoid model and the actual clinical chemotherapeutic efficacy in cholangiocarcinoma patients, assisting in guiding precision medicine and making therapeutic decisions.

Drug sensitivity tests include single drug and drug combination. The organoids that are successfully cultured will be kept in liquid nitrogen for a specific time.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must sign an informed consent form;
2. Age 18-75 years old, both male and female;
3. ECOG performance status score (PS score) 0-2;
4. Child-Pugh score A period;
5. Cholangiocarcinoma with negative margins confirmed by histopathology;
6. Have not received any systemic treatment within 6 months;
7. The functional indicators of important organs meet the following requirements (1)Neutrophils≥1.5*109/L; platelets≥100*109/L; hemoglobin≥9g/dl; serum albumin≥3g/dl; (2)Thyroid-stimulating hormone (TSH) ≤ 2 times the upper limit of normal, and T3 and T4 are in the normal range; (3)Bilirubin ≤ 1.5 times the upper limit of normal; ALT and AST ≤ 3 times the upper limit of normal; (4)Serum creatinine ≤ 1.5 times the upper limit of normal, and creatinine clearance ≥ 60ml/min (calculated by Cockcroft-Gault formula);
8. For women who are not breastfeeding or pregnant, use contraception during treatment or 12 months after the end of treatment.

Exclusion Criteria:

1. Unresectable cholangiocarcinoma patients or postoperative diagnosis of cholangiocarcinoma recurrence and metastasis;
2. Past or simultaneous suffering from other malignant tumors;
3. Have used gemcitabine-based chemotherapy or radiotherapy within 6 months;
4. Severe cardiopulmonary and renal dysfunction;
5. Hypertension that is difficult to control with drugs (systolic blood pressure (BP) ≥140 mmHg and/or diastolic blood pressure ≥90mmHg) (based on the average of ≥3 BP readings obtained by ≥2 measurements);
6. Abnormal coagulation function (PT>14s), have bleeding tendency or are receiving thrombolysis or anticoagulation therapy;
7. After antiviral treatment, HBV DNA>2000 copies/ml, HCV RNA>1000;
8. A history of esophageal and gastric varices, significant clinically significant bleeding symptoms or a clear tendency to appear within 3 months before enrollment;
9. Active infections requiring systemic treatment; patients with active tuberculosis infection within 1 year before enrollment; a history of active tuberculosis infection more than 1 year before enrollment, and no formal anti-tuberculosis treatment or tuberculosis Still in the active period;
10. Human immunodeficiency virus (HIV, HIV1/2 antibody) positive;
11. A history of psychotropic drug abuse, alcohol or drug abuse;
12. Known to have a history of severe allergies to any platinum drugs, or gemcitabine;
13. Other factors judged by the investigator may affect the safety of the subjects or the compliance of the trial. Such as serious diseases (including mental illness) that require combined treatment, serious laboratory abnormalities, or other family or social factors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically confirmed cholangiocarcinoma patients who underwent radical resection and received post-operation adjuvant chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-11-30 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival status of cholangiocarcinoma patients after radical resection | 12 months
  The cholangiocarcinoma patients after radical resection are regularly followed-up for the progression-free survival status.
Drug sensitivity of patient-derived tumor organoids | 2 months
  The drug sensitivity is tested on patient-derived tumor organoids, which is evaluated using Promega CellTiter-Glo 3D Cell Viability Assay to calculate the relative IC50, and is compared with the actual chemotherapeutic efficacy of cholangiocarcinoma patients.

CONTACTS AND LOCATIONS:
Overall Officials: Chao Liu, PhD, Principal Investigator — Department of Biliary and Pancreatic Surgery, Sun Yat-sen Memorial Hospital, Sun Yat-sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No